CLINICAL TRIAL: NCT00505921
Title: Autologous and Allogeneic Transplantation for T-Cell Lymphoma: Impact of Campath -1H and Soluble CD52
Brief Title: Autologous and Allogenic Transplantation With Campath-1H for T-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID02-645
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Lymphoma
Keywords: T-Cell Lymphoma; Lymphoma; Campath-1H; Allogenic Transplantation; Stem Cell Transplant; Alemtuzumab
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell | interventions — Alemtuzumab; Granulocyte Colony-Stimulating Factor; Filgrastim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; sargramostim; Carmustine; Stem Cell Transplantation; Cytarabine; Etoposide; etoposide phosphate; Melphalan; fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath-1H (Experimental): 3 mg in vivo Day 1; 10 mg Day 2; 30 mg Days 3 and 10 of chemotherapy treatment. Transplantation on Day 0.
  Preparative Regimen For Autologous Stem Cell Transplantation: BEAM (BCNU 300 mg/m2 intravenous (IV) over 1 hour on day -6, cytarabine 200 mg/m2 IV twice a day on day -5 through -2 (total 8 doses), etoposide 200 mg/m2 IV twice on day -5 to -2 (total 8 doses), and Melphalan 140 mg/m2 IV on day -1. Beginning on day +5 G-CSF 10 mg/kg sc (in a.m.) and GM-SCF 250 m/m2 on Day +5 (in p.m.)
  Preparative Regimen For Allogenic Stem Cell Transplantation: Campath 15mg/day (days -6 to -4), fludarabine 30 mg/m2 IV/day (days -6 to -4) and cyclophosphamide 750 mg/m2 IV/day (1000 mg/m2 IV/day if unrelated) (days -6 to -4). Low dose total body irradiation of 2 Gy day 0.
  Interventions: Drug: Campath-1H; Drug: G-CSF; Drug: GM-CSF; Drug: BCNU; Drug: Stem Cell Transplant; Drug: Preparative Regimen for Allogenic Stem Cell Transplantation; Drug: Cytarabine; Drug: Etoposide; Drug: Melphalan; Drug: Campath; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Low dose total body irradiation

INTERVENTIONS:
Drug: Campath-1H — 3 mg through the catheter Day 1 then 10 mg on Day 2, and 30 mg on Days 3 and 10 of chemotherapy treatment.
  Other Names: Alemtuzumab; Campath
Drug: G-CSF — 10 mg/kg subcutaneously (sc) on day +5 (in a.m.) for Stem Cell Mobilization.
  Other Names: Granulocyte colony-stimulating factor; GCSF; Filgrastim; Neupogen
Drug: GM-CSF — 250 m/m2 subcutaneously (sc) on Day +5 (in p.m.) for Stem Cell Mobilization.
  Other Names: Granulocyte-Macrophage Colony Stimulating Factor; Sargramostim; Leukine
Drug: BCNU — 300 mg/m2 IV over 1 hour on day -6
  Other Names: Carmustine; BiCNU
Drug: Stem Cell Transplant — Stem cell infusion on Day 0.
  Other Names: SCT
Drug: Preparative Regimen for Allogenic Stem Cell Transplantation — Campath 15mg/day (days -6 to -4), fludarabine 30 mg/m2 IV/day (days -6 to -4) and cyclophosphamide 750 mg/m2 IV/day (1000 mg/m2 IV/day if unrelated) (days -6 to -4). Low dose total body irradiation of 2 Gy on day 0.
Drug: Cytarabine — 200 mg/m2 IV twice a day on day -5 through -2 (total 8 doses),
  Other Names: ARA; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
Drug: Etoposide — 200 mg/m2 IV twice on day -5 to -2 (total 8 doses)
  Other Names: Etoposide phosphate; VePesid
Drug: Melphalan — 140 mg/m2 IV on day -1.
  Other Names: Alkeran
Drug: Campath — 15 mg/day (days -6 to -4) for preparative regimen Allogenic Stem Cell Transplantation
  Other Names: Alemtuzumab; Campath-1H
Drug: Fludarabine — 30 mg/m2 IV/day (days -6 to -4)
  Other Names: Fludarabine monophosphate; Fludara
Drug: Cyclophosphamide — 750 mg/m2 IV/day (1000 mg/m2 IV/day if unrelated) (days -6 to -4).
  Other Names: Cytoxan; Neosar
Radiation: Low dose total body irradiation — Low dose total body irradiation of 2 Gy day 0.
  Other Names: LD-TBI

SUMMARY:
Primary Objectives:

1. To evaluate the role of autologous and allogenic stem cell transplantation with Campath-1H for patients with peripheral T-cell lymphoma (PTCL).
2. To examine the impact of in-vivo purging with Campath -1H pre-autologous stem transplantation for patients with PTCL.
3. To evaluate the impact of soluble CD52 upon in-vivo purging with Campath-1H.
4. To evaluate the role of Campath -1H in the treatment minimal residual disease after autologous transplantation for PTCL.

DETAILED DESCRIPTION:
Campath is a drug that can specifically attack some types of T-cell lymphoma cells.

Before the study begins, you will have a physical exam, including blood (about 2 tablespoons) and urine tests. Women who are able to have children must have a negative blood pregnancy test. Bone marrow samples will be taken. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anaesthetic and a small amount of bone marrow is withdrawn through a large needle. Patients will have a chest x-ray, an EKG (test to measure the electrical activity of the heart), and tests of lung function. Patients whose disease affects the stomach or intestines may have biopsies of these areas.

Treatment will be given in the hospital at M. D. Anderson. You will need to stay in the hospital for about 3 to 4 weeks.

A central venous catheter (plastic tube) will be placed into the large chest vein. The catheter will be left in place throughout treatment. In order to collect stem cells, G-CSF and GM-CSF will be injected under the skin. This will be done twice a day until the collection of stem cells is complete. You will receive Campath -1H through the catheter on Days 1, 2, 3, and 10 of chemotherapy treatment.

The stem cells will be collected from you starting about 10 to 14 days after chemotherapy is given. The collection process is called apheresis. Blood is removed from the your body and the stem cells are frozen for storage. Stem cell collection takes about 3 hours. Between 3 and 5 sessions may be needed to collect enough stem cells. Sessions will be done once a day.

After stem cells are collected, you will receive high dose Carmustine over 1 hour on Day 1. You will receive cytarabine and etoposide twice a day on Days 2 through 5 and melphalan on Day 6.

One day after finishing the chemotherapy, the stem cells that were collected earlier will be infused back into you over about 30 minutes. G-CSF and GM-CSF will be injected until your white blood cell counts returns to normal.

Blood tests (1-2 tablespoons), urine tests, bone marrow sampling, and x-rays will be done as needed to track the effects of the transplant. You will have transfusions of blood and platelets as needed. Blood tests (1-2 tablespoons) will be done daily while you are in the hospital.

You might have to stay in the Houston area for 2 to 4 weeks after the transplant. After that, you will need to return to Houston every 3 months for the first year, then every 6 months for 5 years. Three months after the transplant, bone marrow exams and other tests will be done. If you show evidence of disease, you will receive another cycle of Campath -1H three times a week for 4-12 weeks. Patients will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. The FDA has approved the drugs used in this study. Their use together in this study is investigational. About 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

Nonmyeloablative Allogeneic Transplantation with Campath-1H for T-cell Lymphoma:

Campath is a drug that can specifically attack some types of T-cell lymphoma cells. In addition, it weakens the immune system, therefore helping to prevent the rejection of donor marrow or stem cells.

TBI is designed to damage the DNA (the genetic material of cells) of cancer cells, which may kill the cancer cells.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Fludarabine is designed to make cancer cells less able to repair damaged DNA. This may increase the likelihood of the cells dying.

Before the study begins, you will have a physical exam, including blood (about 1-2 tablespoons) and urine tests. Women who are able to have children must have a negative blood pregnancy test. Bone marrow samples will be taken. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anaesthetic and a small amount of bone marrow is withdrawn through a large needle. You will have a chest x-ray, CT scans, an EKG (test to measure the electrical activity of the heart), and tests of lung function.

Blood tests (1-2 tablespoons), urine tests, bone marrow sampling, and x-rays will be done as needed to track the effects of the transplant. Patients will have transfusions of blood and platelets as needed. Blood tests (1-2 tablespoons) will be done daily while you are in the hospital.

Campath-1 H will be injected into your vein. This will be done 3 days in a row (Days 1 to 3). The drugs diphenhydramine (Benadryl), acetaminophen (Tylenol) and hydrocortisone will be given in to decrease the risk of or ease side effects.

You will also receive fludarabine and cyclophosphamide daily for 3 days. They will be given starting day of Campath -1H.

All of the chemotherapy drugs will be given through a catheter (plastic tube) that extends into the large chest vein. The catheter will be left in place throughout treatment. After completion of chemotherapy, you will receive TBI, and later on the same day, blood stem cells from a donor will be given through the catheter. G-CSF and GM-CSF, growth factors that promote the production of blood cells, will be injected under the skin once a day until the neutrophil counts recover in the blood.

Tacrolimus will be infused through the vein, starting 2 days before transplant to decrease the risk of graft-versus-host disease. It will be changed to pills after you are discharged from the hospital. For the same purpose, methotrexate will also be given through the vein on Days 1, 3, 6 (and Day 11 if unrelated donor).

Treatment will be given in the hospital at UTMDACC. You will need to stay in the hospital for about 3 to 4 weeks.

You must stay in the Houston area for about 100 days after the transplant. After that, you will need to return to Houston every three months for the first year, then every 6 months for 5 years for blood tests (1-2 tablespoons), urine tests, and CT scans. Bone marrow aspirations and biopsies will also be performed. Patients will be taken off study if the intolerable side effects occur.

This is an investigational study. The FDA has approved the drugs used in this study. Their use together in this study is investigational. About 30 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be less then 70 years old.
* Patients must have chemosensitive disease, having undergone at least partial remission with less then 10% marrow involvement by gross pathologic examination if autologous transplantation is considered.
* Newly diagnosed patients are eligible for autologous transplant. Patients in relapse would receive a non-myeloablative transplant if a sibling donor is available. Otherwise, patients would undergo autologous transplant if International Prognostic Index (IPI) is 0-1, or unrelated transplant if IPI is > 1.

Exclusion Criteria:

* Criteria for exclusion are Human immunodeficiency virus (HIV) or Human T-lymphotropic virus (HTLV) seropositivity, pregnancy, cardiac ejection fraction by echo-cardiogram less than 40%, active central nervous system involvement, serum creatinine greater than 1.6 mg/dl or serum bilirubin greater than 1.5 mg/dl unless due to tumor, Absolute neutrophil count (ANC) less than 1,000/mm3 and platelets less than 100,000/mm3 unless due to tumor, performance status (ECOG scale) greater than 2, pulmonary function test- diffusing capacity of the Lung for Carbon Monoxide (DLCO) less than 40% of predicted, and severe concomitant medical or psychiatric illnesses.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 3/11/2003 to 10/27/2009. All participants were registered at UT MD Anderson Cancer Center
Pre-assignment Details: Eight patients of those twenty-seven registered failed to mobilize an adequate number of stem cells for an autologous transplant and were taken off the study.
Period: Overall Study
Arm/Group | Campath-1H
Started | 27
Completed | 18
Not Completed | 9
Not completed — Ineligible | 1
Not completed — Failed to Mobilize | 8

BASELINE CHARACTERISTICS:
Arm/Group | Campath-1H
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 44 (0) [22 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Participant Progression Free Survival at 2 Years
Description: Progression-free survival defined as the number of participants without evidence of progression or death after 2 years from stem cell transplant.
Time Frame: 2 years
Population: Analysis was per protocol. Nine participants were not eligible for treatment therefore were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Campath-1H
Number analyzed (Participants) | 18
participants | 15

ADVERSE EVENTS:
Time Frame: 5 years and 8 months
Arm/Group | Campath-1H
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-1H (N=18)
hypertension (Cardiac disorders) | 1 (1)
low blood pressure (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
fatigue (Infections and infestations) | 1 (1)
fevers (Infections and infestations) | 3 (3)
Flu-like symptoms-other (General disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 9 (9)
nausea (Gastrointestinal disorders) | 15 (16)
Esophagitis (Gastrointestinal disorders) | 11 (12)
abdominal pain (Gastrointestinal disorders) | 1 (1)
increased creatinine (Renal and urinary disorders) | 5 (5)
cystitis (Renal and urinary disorders) | 1 (1)
Hepatic Alkaine Phos (Hepatobiliary disorders) | 4 (4)
ALT- Transaminase (Hepatobiliary disorders) | 1 (1)
AST-Tranaminase (Hepatobiliary disorders) | 1 (1)
increased bilirubin (Hepatobiliary disorders) | 2 (2)
neutropenia infection (Infections and infestations) | 3 (3)
infection (Infections and infestations) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
involuntary movement (Nervous system disorders) | 1 (1)
neurological other complaints (Nervous system disorders) | 3 (3)
insomnia (General disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Early termination due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No